CLINICAL TRIAL: NCT02948803
Title: A Smartphone-based Intervention to Promote an Active Lifestyle in Low Educated Working Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11U8114N
Record Dates: First submitted 2016-10-06; First posted 2016-10-28 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Physical Activity
Keywords: intervention; mHealth; physical activity; active transport; smartphone; application
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: pre, post, follow up measurements with an intervention and control group

ARMS (2):
- Intervention group (Experimental): smartphone based intervention with Active Coach app: participants in the intervention group will use a newly developed smartphone app in combination with a Fitbit Charge activity tracker for 9 weeks. The app aims to promote an active lifestyle.
  Interventions: Behavioral: smartphone based intervention with Active Coach app
- control group (No Intervention): participants in the control groups only receive a flyer with standard information about an active lifestyle

INTERVENTIONS:
Behavioral: smartphone based intervention with Active Coach app
  Arms: Intervention group

SUMMARY:
The aim of this smartphone-based intervention study is to determine whether a newly developed app is effective in promoting an active lifestyle in low educated working young adults.

DETAILED DESCRIPTION:
A stepwise approach was used to develop a new native Android smartphone app (Active Coach). This app aims to promote an active lifestyle (through physical activity and active transport) in low educated working young adults. The development of this app is based on theory, evidence and user's experiences. The app focuses on four determinants (knowledge, attitude (perceived benefits and perceived barriers), social support and self-efficacy) and includes several behavioral change techniques (self-monitoring, goal-setting, feedback on behavior, review behavior goals, instruction on how to perform the behavior, information about health consequences, enhancing network linkages and prompts/cues). Furthermore, the app works in combinations with a wearable activity tracker (Fitbit Charge) to track users activity behavior.

For the smartphone-based intervention, 120 low educated working young adults are being recruited via purposeful convenience sampling though companies and employers. Participants can not have any medical conditions that prevent them from being physically active and they need to own an Android smartphone. Fitbit Charge activity trackers will be provided. The participants will be randomly divided in the intervention group or the standard information control group. The intervention period will be nine weeks. At the beginning and the end of the intervention period, physical activity levels will be objectively measured with accelerometers. Follow-up measurements will be conducted 12 weeks after the end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 28 years old
* low educated (maximum secondary school, no higher education (university or college)
* employed
* dutch speaking
* owning an Android smartphone

Exclusion Criteria:

* being very physically active (already reaching the recommended 30 minutes of physical activity a day)

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-17 (Actual)

PRIMARY OUTCOMES:
change in physical activity: objective | The outcome will be measured at baseline (before start intervention), posttest (9 weeks after the start of the intervention) and follow-up (12 weeks after the posttest)
  physical activity will be objectively measured by accelerometers (Actigraph)
change in physical activity: self-reported | The outcome will be measured at baseline (before start intervention), posttest (9 weeks after the start of the intervention) and follow-up (12 weeks after the posttest)
  physical activity will be measured via the International Physical Activity Questionnaire (IPAQ, long version)

SECONDARY OUTCOMES:
Change in perceived benefits towards physical activity and active transport | The outcome will be measured at baseline (before start intervention), posttest (9 weeks after the start of the intervention) and follow-up (12 weeks after the posttest)
  benefits will be measured via fifteen items with a five-point answer format
Change in perceived barriers towards physical activity and active transport | The outcome will be measured at baseline (before start intervention), posttest (9 weeks after the start of the intervention) and follow-up (12 weeks after the posttest)
  barriers will be measured via fifteen items with a five-point answer format
Change in social support towards physical activity and active transport | The outcome will be measured at baseline (before start intervention), posttest (9 weeks after the start of the intervention) and follow-up (12 weeks after the posttest)
  social support will be measured via nine items with a five-point answer format
Change in self-efficacy towards physical activity and active transport | The outcome will be measured at baseline (before start intervention), posttest (9 weeks after the start of the intervention) and follow-up (12 weeks after the posttest)
  self-efficacy will be measured via eight items with a five-point answer format
Change in knowledge towards physical activity and active transport | The outcome will be measured at baseline (before start intervention), posttest (9 weeks after the start of the intervention) and follow-up (12 weeks after the posttest)
  knowledge will be measured via one item with a six-point answer format

CONTACTS AND LOCATIONS:
Overall Officials: Dorien Simons, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simons D, De Bourdeaudhuij I, Clarys P, De Cocker K, Vandelanotte C, Deforche B. Effect and Process Evaluation of a Smartphone App to Promote an Active Lifestyle in Lower Educated Working Young Adults: Cluster Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Aug 24;6(8):e10003. doi: 10.2196/10003. PMID 30143477